CLINICAL TRIAL: NCT01658852
Title: Effects and Safety of Metronidazole in Patients With Gastrectomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of difficulties on recruiting participants
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myung-gui Choi, prof., The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gastrectomy-MDZ-001
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Post Gastrectomy State
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Metronidazole (Active Comparator): active drug: metronidazole 500mg three time per day for 10 days
  Interventions: Drug: metronidazole
- Placebo (Placebo Comparator): Placebo three times per day for 10days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metronidazole
  Arms: Metronidazole
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recent study showed that SIBO is common among postgastrectomy patients and It appears to be associated with postprandial intestinal symptoms and might aggravate late hypoglycemia. SIBO could be a new therapeutic target for managing intestinal symptoms in postgastrectomy patients.The purpose of this study is to determine whether antiboitic (metronidazole) is effective in patients with postgasrectomy syndrome

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70
* gastrectomy for early gastric cancer with complete resection
* no reccurrence after follow up more than 6 months
* identified small bowel bacterial overgrowth by hydrogen breath test
* symptoms of postgastrectomy syndrome

Exclusion Criteria:

* hypersensive to metronidazole
* systemic chemotherapy history
* other organic gastrointestinal disease (inflammatory bowel disease, carcinoid syndrome, amyloidosis, intestinal obstruction)
* other gastrointestinal operation history except appendectomy, cholecystectomy)
* recent colonoscopic examination (within 30 days)
* uncontrolled psychopathy
* drug or alcohol abuser
* pregnant or breast feeding woman
* recent history of antibiotics treatment (within 90 days)
* recent history of PPI or H2 blocker treatment (within 30 dyas)
* recent history of probiotics treatment (within 30 dyas)
* recent history of prokinetics or antispasmotic treatment (within 15 days)
* severe systemic illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Patient's Global Assessment of abdominal symptom | 4 week